CLINICAL TRIAL: NCT06351176
Title: Impact of Glycemic Control on Skeletal Outcomes in Adults With Type 1 Diabetes : DenSiFy (Diabetes Spine Fractures) Cohort
Brief Title: Impact of Glycemic Control on Skeletal Outcomes in Adults With Type 1 Diabetes
Acronym: DenSiFy cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Claudia Gagnon, MD, CHU de Quebec-Universite Laval
Other Study IDs: 2024-6819
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 1; Bone Health; Bone Loss; Bone Diseases, Metabolic; Hyperglycaemia Due to Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Bone Diseases, Metabolic | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with type 1 diabetes
  Interventions: Diagnostic Test: Clinical tests; Diagnostic Test: Biochemical tests; Diagnostic Test: DXA scan with TBS and VFA; Diagnostic Test: AGEReader
- Healthy controls
  Interventions: Diagnostic Test: Clinical tests; Diagnostic Test: Biochemical tests; Diagnostic Test: DXA scan with TBS and VFA; Diagnostic Test: AGEReader

INTERVENTIONS:
Diagnostic Test: Clinical tests — The investigators perform the following clinical tests: vibration threshold test, monofilament test, and height, weight and waist circumference measurement in every participant.
Diagnostic Test: Biochemical tests — The investigators perform blood and urine tests in every participant.
Diagnostic Test: DXA scan with TBS and VFA — The investigators perform a dual energy x-ray absorptiometry (DXA scan or osteodensitometry) including trabecular bone score (TBS) and Vertebral Fracture Assessment (VFA) in every participant.
Diagnostic Test: AGEReader — The investigators perform a skin advanced glycation end products (AGEs) measurement with the AGE Reader machine in every participant.

SUMMARY:
Background : Type 1 diabetes (T1D) is associated with an increased risk of fractures. The mechanisms accounting for this bone fragility are not yet fully understood. As T1D is often diagnosed in childhood or early adulthood, the lower bone mineral density (BMD) and deteriorated bone microarchitecture observed in T1D may reflect changes in the bone that occurred before or at the time of peak bone mass achievement. There is a lack of high-quality prospective studies to determine whether adults with T1D continue to lose BMD or deteriorate bone quality compared with controls. Moreover, while chronic hyperglycemia is a risk factor for fracture in T1D, it is unknown if better glycemic control affects bone outcomes.

This prospective multicenter cohort study aims: (1) To compare the changes in the following outcomes over 4 years in adults with T1D and controls without diabetes of similar age, sex and body-mass index distribution: BMD by dual-energy X-ray absorptiometry (DXA) at the femoral neck, hip, spine, and radius, trabecular bone score (TBS) by DXA, and serum biochemical markers of bone turnover (BTMs); (2) To evaluate whether long-term glycemic control or the presence of a microvascular complication are independent predictors of the changes in BMD and TBS in people with T1D.

ELIGIBILITY:
Individuals with type 1 diabetes who have participated in the DenSiFy (Diabetes Spine Fractures) study (NCT04064437)

Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least 5 years;
* Age 20 years and older.

Exclusion Criteria:

* Pregnancy, delivery or breastfeeding in the past 6 months;
* Conditions associated with bone disease (significant liver disease, intestinal malabsorption other than celiac disease, organ transplant, active cancer, rheumatoid arthritis, hyperthyroidism, hypothyroidism with abnormal TSH, hyperparathyroidism, hypoparathyroidism, hypogonadism, acromegaly, Cushing syndrome, adrenal insufficiency);
* Any of these medications since the first DenSiFy study visit : biphosphonates, teriparatide, denosumab, calcitonin, glucocorticoids ≥ 7,5 mg prednisone/day or equivalency ≥ 3 months, aromatase inhibitors, antiandrogens, antiepileptic drugs, anticoagulants, thiazolidinediones;
* Inability to consent.

Healthy controls who have participated in the DenSiFy (Diabetes Spine Fractures) study (NCT04064437)

Inclusion Criteria:

* Age 20 years and older.

Exclusion Criteria :

* As above (as individuals with diabetes), and :
* Diagnosis of diabetes or prediabetes;
* Celiac disease;
* Chronic kidney disease (CrCl < 60 mL/min).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 127 individuals with type 1 diabetes and 65 healthy subjects from the DenSiFy (Diabetes Spine Fractures) study (NCT04064437)
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Change in areal bone mineral density (aBMD) at the femoral neck in g/cm2 | Between the baseline and the 4-year visit
  aBMD measured by DXA scan

SECONDARY OUTCOMES:
Change in areal bone mineral density (aBMD) at the spine in g/cm2 | Between the baseline and the 4-year visit
  aBMD measured by DXA scan
Change in areal bone mineral density (aBMD) at the total hip in g/cm2 | Between the baseline and the 4-year visit
  aBMD measured by DXA scan
Change in areal bone mineral density (aBMD) at the distal third of radius in g/cm2 | Between the baseline and the 4-year visit
  aBMD measured by DXA scan
Change in Trabecular bone score (TBS) (unitless) | Between the baseline and the 4-year visit
  TBS with the software TBSinSight
Glycemic control, assessed with mean glycated hemoglobin (HbA1c) of the past 7 years | 4-year visit
  Mean HbA1c of the past 7 years from all the available HbA1c in the medical record
Glycemic control, assessed with skin advanced glycation end products (AGEs) | 4-year visit
  Skin AGEs measured with AGEReader (autofluorescence)
Presence of a microvascular complication (neuropathy, nephropathy, retinopathy) | 4-year visit
  From the information available in the medical record and from monofilament and vibration testing (for neuropathy) and from microalbuminuria (nephropathy)

OTHER OUTCOMES:
Areal bone mineral density at the femoral neck, g/cm2 | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the femoral neck, T-Score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the femoral neck, Z-Score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the total hip, g/cm2 | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the total hip, T-score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the total hip, Z-score | 4 year visit
  Measured by DXA scan
Areal bone mineral density at the spine, g/cm2 | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the spine, T-Score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the spine, Z-score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the distal third of radius, g/cm2 | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the distal third of radius, T-score | 4-year visit
  Measured by DXA scan
Areal bone mineral density at the distal third of radius, Z-score | 4-year visit
  Measured by DXA scan
Trabecular bone score (TBS) at the lumbar spine (L1-L4) (unitless) | 4-year visit
  TBS calculated with the software TBSinSight
Vertebral Fracture Assessment (VFA) from the T4 to L5 vertebrae to detect the presence of vertebral fracture | 4-year visit
  Image acquired by DXA
Lean mass (arm, leg, trunk, android, gynoid and total) (g) | 4-year visit
  Body composition measured by DXA scan
Fat mass (arm, leg, trunk, android, gynoid and total) (g) | 4-year visit
  Body composition measured by DXA scan
C-terminal cross-linking telopeptide of type I collagen (C-telopeptide, CTX) (ng/mL) | 4-year visit
  Bone turnover marker, bone resorption (serum)
Procollagen type 1 N-terminal propeptide (P1NP) (ng/mL) | 4-year visit
  Bone turnover marker, bone formation (serum)
Osteocalcin (ng/mL) | 4-year visit
  Bone turnover marker, bone formation (serum)
Sclerostin (pmol/mL) | 4-year visit
  Inhibitor of bone formation (serum)
Change in C-terminal cross-linking telopeptide of type I collagen (C-telopeptide, CTX) (ng/mL) | Between the baseline and the 4-year visit
  Bone turnover marker, bone resorption (serum)
Change in osteocalcin (ng/mL) | Between the baseline and the 4-year visit
  Bone turnover marker, bone formation (serum)
Change in procollagen type 1 N-terminal propeptide (P1NP) (ng/mL) | Between the baseline and the 4-year visit
  Bone turnover marker, bone formation (serum)
Change in sclerostin (pmol/mL) | Between the baseline and the 4-year visit
  Inhibitor of bone formation (serum)
Skin advanced glycation end-products (AGEs) (arbitrary units) | 4-year visit
  Measured with AGEReader (autofluorescence)
Glycated hemoglobin (HbA1c, %) | 4-year visit
  Diabetes control marker
Fasting glucose (mmol/L) | 4-year visit
  Blood level measurement
Complete blood count | 4-year visit
  Blood level measurement
Thyroid-stimulating hormone (TSH) (mU/L) | 4-year visit
  Blood level measurement
Lipid panel (total cholesterol, LDL-cholesterol, HDL-cholesterol, non-HDL-cholesterol, total cholesterol/HDL-cholesterol ratio, triglycerides, in mmol/L) | 4-year visit
  Blood level measurement
Creatinine (umol/L) | 4-year visit
  Blood level measurement
Microalbuminuria (mg/mmol) | 4-year visit
  Urine microalbuminuria/ urine creatinine ratio measurement
Liver enzymes (AST, ALT) (U/L) | 4-year visit
  Blood level measurement
Calcium (mmol/L) | 4-year visit
  Blood level measurement
Albumine (g/L) | 4-year visit
  Blood level measurement
Phosphate (mmol/L) | 4-year visit
  Blood level measurement
25-hydroxyvitamin D3 (nmol/L) | 4-year visit
  Blood level measurement
Parathormone (PTH) (ng/L) | 4-year visit
  Blood level measurement
Antitransglutaminase antibodies (U/mL) | 4-year visit
  Blood level measurement
Immunoglobulin A (IgA) (g/L) | 4-year visit
  Blood level measurement
Insulin like growth factor-1 (IGF-1) (ng/mL) | 4-year visit
  Blood level measurement
Follicle stimulating hormone (FSH, women) (U/L) | 4-year visit
  Blood level measurement
Total testosterone (men) (nmol/L) | 4-year visit
  Blood level measurement
Sex hormone-binding globulin (SHBG, men) (nmol/L) | 4-year visit
  Blood level measurement

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, MD, Principal Investigator — CHU de Québec- Université Laval
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal (IRCM), Montreal, Quebec
  - Centre de recherche du CHU de Québec-Université Laval, Québec, Quebec